CLINICAL TRIAL: NCT03751163
Title: Randomized, Controlled, Double-blind Study of Oral Tranexamic Acid and Topical Hydroquinone in the Treatment of Melasma
Brief Title: Oral Tranexamic Acid and Topical Hydroquinone in the Treatment of Melasma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Nahla Shihab, Principal Investigator, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 008
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Melasma
Keywords: melasma; tranexamic acid; hydroquinone; mMASI; mexameter
MeSH Terms: conditions — Melanosis | interventions — hydroquinone; Sunscreening Agents; Sun Protection Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Active Comparator): Tranexamic acid 250 mg po bid 12 weeks 4% Hydroquinone cream qhs 12 weeks sunscreen spf 30 qam 24 weeks
  Interventions: Drug: Tranexamic Acid Oral Product; Drug: Hydroquinone 4% Cream; Other: Sunscreen
- Control (Placebo Comparator): Placebo po bid 12 weeks 4% Hydroquinone cream qhs 12 weeks sunscreen spf 30 qam 24 weeks
  Interventions: Drug: Hydroquinone 4% Cream; Other: Sunscreen; Device: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid Oral Product — Encapsulated tranexamic acid 250 mg
  Other Names: TA
  Arms: Study
Drug: Hydroquinone 4% Cream — Hydroquinone 4% Cream
  Other Names: HQ
Other: Sunscreen — Sunscreen SPF 30
  Other Names: Sun Protection
Device: Placebo — Encapsulated placebo
  Arms: Control

SUMMARY:
This study assess the effectiveness of oral tranexamic acid in combination with hydroquinone cream in the treatment of melasma.

DETAILED DESCRIPTION:
Hydroquinone (HQ) is considered the gold standard depigmenting agent for melasma, nevertheless, many patients are recalcitrant to this treatment.

Recent studies have shown that tranexamic acid, a plasmin inhibitor, can prevent UV-induced pigmentation.

ELIGIBILITY:
Inclusion Criteria:

* moderate melasma (subject with mMASI score of 5 to 7.9),
* severe melasma (subject with mMASI score ≥ 8),
* willing to follow up for 6 months.

Exclusion Criteria:

* pregnant women,
* nursing women,
* women on exogenous hormones
* current treatment with blood thinners,
* had a history of thrombosis,
* had an abnormal kidney function,
* use of topical hydroquinone within 3 months of study enrollment,
* use of topical steroids, vitamin A analogs, chemical peels within 1 month of study

Ages: 21 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2017-04-02 (Actual); Study Completion 2017-04-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline mMASI Score at week 12 | Baseline, week 2, 12, 24
  modified Melasma Area and Severity Index (mMASI) score was performed by rating darkness and area of involvement of 4 areas of the face (forehead, right malar, left malar, chin)
  Scoring system: A, Area of involvement rated 0 to 6: 0 indicates absent;
  1, <10%; 2, 10% to 29%; 3, 30% to 49%; 4, 50% to 69%; 5, 70% to 89%; 6, 90% to 100%. D, Darkness rated 0 to 4: 0 indicates absent; 1, slight; 2, mild; 3, marked; 4, severe. b Total mMASI score range is 0 to 24 and calculated by adding scores for 4 areas of the face.
  Forehead (0.3xAxD) + Right Malar (0.3xAxD) + Left Malar (0.3xAxD) + Chin (0.1xAxD)

SECONDARY OUTCOMES:
Melanin index | Baseline, week 2, 12, 24
  difference in pigmentation readings between involved and adjacent uninvolved skin, was measured using a mexameter.
  Mexameter is a simple, rapid, and completely non-invasive instrument which measures skin pigmentation. The device has a probe which is gently pressed on the skin and painlessly records the level of pigmentation using a range of 1-1000, with 1 corresponding to white and 1000 to black.